CLINICAL TRIAL: NCT05509491
Title: Postural Awareness Program With Exercises In Patients With Neck Pain
Brief Title: Effectiveness of A Telehealth Postural Awareness Program Combined With Exercise In People With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Director, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-191
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Neck Pain
Keywords: neck pain; neck; telehealth; awareness; posture; exercise
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 12-week physiotherapist delivered a postural awareness program with exercises
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postural Awareness Program with Exercises in people with neck pain (Experimental): Postural education, bad posture, good posture, awareness, their effects in daily life
  Interventions: Behavioral: A postural awareness program with exercises

INTERVENTIONS:
Behavioral: A postural awareness program with exercises — A program about postural awareness, bad posture, good posture and their effects on daily life

SUMMARY:
People with neck pain often experience pain, neck disability, and poor quality of life. Postural-based awareness programs are evidence-based interventions for postural problems and neck pain disorders. This study aims to determine the effectiveness of a telehealth physiotherapist-delivered postural awareness program combined with exercise in people with neck pain. Pain, neck disability, leisure time management, and exercise stage of change were evaluated.

DETAILED DESCRIPTION:
Pain with visual analog scale, neck disability with Neck Disability Index, Leisure time management with Leisure Time Management Scale, and exercise stage of change with exercise Stage of change Scale were determined. The authors aim to find out if there are any changes before and after the program on the pain, neck disability, and evaluation subscale of the leisure time management scale, and exercise stage of change of participants.

ELIGIBILITY:
Inclusion Criteria:

* being aged 18 years or over,
* volunteering to take part in the study,
* being a student of online education,
* without a history of any neurological or orthopedic problem,
* with resting neck pain (as measured by the VAS) lasting ≤30 days
* that is aggravated by movement without extending distal to the shoulders.

Exclusion Criteria:

* rheumatological diseases, malignity or structural deformities,
* previous surgical intervention related to the neck region,
* severe pain (more than 7 in 0 to 10 VAS)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Neck pain | 5 minute
  Visual Analog Scale- The evaluations of this study was performed at beginning and end of study. Neck pain was determined with Visual Analog Scale with 0 indicating "no pain", 10 indicating "the most severe pain

SECONDARY OUTCOMES:
Neck Disability | 10 minute
  Neck Disability Index-The Neck Disability Index consists of 10 items: pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping and recreation. Individuals included in the study were asked to rate each title between 0 (no disability) and 5 (complete disability). The total score ranges between 0 (no disability) and 50 (complete disability)
Leisure Time Management | 10 minute
  Leisure Time Management- This scale consists of four sub-dimensions and 15 items. These sub-dimensions were investigated as "evaluation", "programming", "leisure attitude", "goal setting and method". The answer codes of each item vary between 1 and 5 as a Likert type.
Exercise Stage of Change | 10 minute
  Exercise Stage of Change Scale-The "Exercise Behavior Change Steps Questionnaire" aims to determine the individual's exercise behavior steps. The four items in the questionnaire, in which the participants' wishes for exercise are tried to be determined, are answered as yes/no. Individuals' intention to exercise and their habits of participating in exercise are divided into five different exercise behavior steps according to their responses to the items: Pre-tendency, Tendency, Preparation, Movement and Continuity.

CONTACTS AND LOCATIONS:
Overall Officials: Tezel Y Şahan, pHD, Study Chair — University of Health science
Locations (1):
- Tezel Yıldırım Şahan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The authors decided that if a researcher want ıpd than they will send them with e mail

REFERENCES:
- [Background] Bennell KL, Jones SE, Hinman RS, McManus F, Lamb KE, Quicke JG, Sumithran P, Prendergast J, George ES, Holden MA, Foster NE, Allison K. Effectiveness of a telehealth physiotherapist-delivered intensive dietary weight loss program combined with exercise in people with knee osteoarthritis and overweight or obesity: study protocol for the POWER randomized controlled trial. BMC Musculoskelet Disord. 2022 Jul 30;23(1):733. doi: 10.1186/s12891-022-05685-z. PMID 35907828
- [Background] Alfawaz S, Lohman E, Alameri M, Daher N, Jaber H. Effect of adding stretching to standardized procedures on cervical range of motion, pain, and disability in patients with non-specific mechanical neck pain: A randomized clinical trial. J Bodyw Mov Ther. 2020 Jul;24(3):50-58. doi: 10.1016/j.jbmt.2020.02.020. Epub 2020 Feb 22. PMID 32826008
- [Background] Toprak Celenay S, Mete O, Sari A, Ozer Kaya D. A comparison of kinesio taping and classical massage in addition to cervical stabilization exercise in patients with chronic neck pain. Complement Ther Clin Pract. 2021 May;43:101381. doi: 10.1016/j.ctcp.2021.101381. Epub 2021 Apr 2. PMID 33831805
- [Background] Lauche R, Wayne PM, Fehr J, Stumpe C, Dobos G, Cramer H. Does Postural Awareness Contribute to Exercise-Induced Improvements in Neck Pain Intensity? A Secondary Analysis of a Randomized Controlled Trial Evaluating Tai Chi and Neck Exercises. Spine (Phila Pa 1976). 2017 Aug 15;42(16):1195-1200. doi: 10.1097/BRS.0000000000002078. PMID 28146026